CLINICAL TRIAL: NCT01028677
Title: Oxytocin Treatment of Social Deficits and Paranoia in Schizophrenia
Brief Title: Oxytocin Treatment of Schizophrenia
Acronym: OTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Cort Pedersen, MD, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-0879
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Paranoia; Schizophrenia; Schizoaffective Disorder
Keywords: oxytocin; social cognition; social skill; social functioning; paranoia; psychotic symptoms; schizophrenia; social deficits; intranasal administration
MeSH Terms: conditions — Paranoid Disorders; Schizophrenia; Psychotic Disorders; Social Skills; Social Adjustment | interventions — Oxytocin; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intranasal spray with oxytocin (Experimental): Twice daily intranasal oxytocin spray (24 IU, 6 insufflations/dose) for 6 weeks
  Interventions: Drug: intranasal spray with oxytocin
- intranasal spray without oxytocin (Placebo Comparator): Twice daily intranasal spray without oxytocin (six 0.1 ml insufflations/dose) for 6 weeks.
  Interventions: Other: nasal spray without oxytocin

INTERVENTIONS:
Drug: intranasal spray with oxytocin — 6 insufflations (24 IU of oxytocin total) given twice daily for 6 weeks
  Other Names: Syntocinon Spray
  Arms: intranasal spray with oxytocin
Other: nasal spray without oxytocin — 6 insufflations of nasal spray without oxytocin (0.1 metered dose/insufflation) twice daily for 6 weeks
  Arms: intranasal spray without oxytocin

SUMMARY:
Purpose: Test whether intranasal administration of the neuropeptide, oxytocin, improves social cognition, social functioning and decreases paranoia and other psychotic symptoms in schizophrenia.

Participants: Up to 80 adults with schizophrenia for at least one year and with a high rating for paranoia.

Procedures (methods): Oxytocin or placebo will be administered twice daily in an intranasal spray (6 insufflations/dose or 24 IU) for 6 weeks. Before, during and at the end of the trial, each subject will undergo social cognitive measures (primary outcomes) and psychiatric symptom ratings (secondary outcomes).

DETAILED DESCRIPTION:
Inclusion criteria: meeting Diagnostic and Statistical Manual IV (DSM-IV) criteria for paranoid or undifferentiated schizophrenia for at least 1 year; scoring > 4 on the suspiciousness/persecution (hereafter referred to as paranoia) subscale of the Positive and Negative Symptom Scale (PANSS) or 3 on the paranoia subscale and > 3 on the hostility, active social avoidance, passive/apathetic social withdrawal or uncooperativeness subscale and > 60 on the full PANSS: stability of symptom severity and on the same medication(s) and dose(s) for at least 1 month; low to moderate depressive symptoms.

Exclusion criteria: low literacy as indicated by an inability to read and understand the consent form; dependence on substances other than tobacco or caffeine; positive urine drug screen for illegal substances or drugs that have not been prescribed; debilitating medical conditions (including AIDS; HIV infection alone will not be grounds for exclusion); major surgery or trauma in the past year will be grounds for exclusion although subjects determined to be recovered and stable may be included at the discretion of the Principal Investigator (PI); pregnancy, breast-feeding; having given birth in the past 6 months or breast-feeding in the past 3 months. Individuals judged unable to learn self-administration of intranasal treatments and/or not sufficiently reliable to do so will be excluded. Abnormalities found during medical evaluation will be grounds for exclusion (see details below) although subjects with laboratory measures somewhat out of the normal range may be included at the discretion of Drs. Pedersen, Gilmore, Rau and/or Salimi.

Study Design: Randomized, double-blind, placebo-controlled design. Up to 80 subjects will complete the protocol: 40 will receive oxytocin; 40 placebo. Prior to the treatment trial, baseline measures will be obtained. Social cognition and psychiatric symptoms will be measured at Baseline and at 6 weeks of the 6 week treatment trial.

Procedures: Subjects will be recruited from the University of North Carolina (UNC) Department of Psychiatry outpatient clinics and the community. If total Positive and Negative Symptoms Scale (PANSS) score is > or equal to 60, PANSS sub-score for suspiciousness/persecution is > or equal to 4, their medical history will be reviewed including medications and dosages over the past month. If they do not have exclusionary medical or medication history, their psychiatric history will be reviewed. If necessary to confirm their diagnosis, they will undergo the Structured Clinical Interview for DSM-IV (SCID) patient version. If they have met criteria for schizophrenia, paranoid or undifferentiated type, for at least one year, they will undergo a physical exam and blood will be drawn and urine collected for laboratory measures including complete blooc count (CBC), electrolytes, blood urea nitrogen (BUN), creatinine, liver function tests, glucose, thyroid-stimulating hormone (TSH), urinanalysis, urine drug screen and pregnancy test. This initial evaluation may require up to 3-4 hours. Prospective subjects will be encouraged to rest for 20-30 minutes between the initial interviews (PANSS, SCID) and the history, physical exam and blood/urine collections. Psychiatric, medical and medication history will be confirmed by reviewing medical records and contacting clinicians in charge of the prospective subject's psychiatric care. The initial evaluation will be conducted in the Clinical and Translational Research Center (CTRC) outpatient clinic or at the UNC Psychiatry Clinical Research Unit (CRU) at Central Regional Hospital (Raleigh or Butner).

SCID, PANSS, other psychological results and medical labs and history will be reviewed during conferences with Dr. Pedersen accompanied by Drs. Gilmore, Salimi and/or Rau. Consensus decisions will be made during these conferences about whether subjects meet the diagnostic and other criteria for inclusion in the study.

For subjects who meet study criteria, baseline measurements of social cognition, social competence, social functioning, paranoia, other psychotic and psychiatric symptoms will be obtained.

During the treatment trial, twice daily test treatments will be self-administered by subjects in the morning shortly after breakfast and late in the afternoon/early evening prior to dinner. Each treatment will consist of 6 insufflations (3/nostril alternating between nostrils) of Syntocinon Spray (Novartis), which contains approximately 24 international units (IU) of oxytocin, or placebo. There will be a 30-60 second pause between each insufflation. The placebo solution will be a solution that has all ingredients in Syntocinon Spray except for oxytocin in 2 oz vials containing 30 ml of solution designed to deliver 0.1 ml metered volume per insufflation. Treatment assignments will be random within each gender.

Social cognition and competence testing will begin 50 min after the morning treatment at 6 weeks (day 42) of the treatment trial and will be followed by ratings of psychotic, mood and anxiety symptoms (requiring 1-3 hr depending on how much social cognition testing is done). The Emotion Recognition-40, Reading the Mind in the Eyes test (Eyes Test), Interpersonal Reactivity Index and Trustworthiness Tasks, Brune Theory of Mind Task, as well as psychiatric ratings will be conducted at all time points.

Participants will be trained by research nurses during their first dosing with test substance in intranasal self-administration shortly after baseline measurements are completed. They will also be given written instructions about the timing of each day's test treatments and other procedures to follow at home. They will be given one 2 ounce vial containing 30 ml of test substance to last until their first outpatient clinic testing appointment and instructed when to begin the twice daily intranasal treatments. They will self administer test substance at the site so staff can confirm they are using proper technique. In addition to social cognition/competence testing and psychiatric ratings, blood samples as well as vital signs will be obtained during these visits. At 40 min after the last intranasal insufflation, blood (15 ml) will be drawn to measure plasma oxytocin concentrations and other lab values (sodium, potassium, glucose [treatment day 42], CBC, BUN, creatinine, liver function tests [treatment days 42]). An electrocardiogram (ECG) will also be obtained on the morning of treatment days 42 approximately 3-4 hr after intranasal treatment (when social cognition/competence testing and psychiatric ratings are completed). Urine will also be collected from female subjects on the day of baseline measurements and on treatment day 42 for pregnancy testing. These same procedures will conducted on the morning of treatment day 42 in participants studied as inpatients.

After procedures at the study site on the morning of treatment days 14 and 28, outpatient subjects will be given a new vial containing 30 ml test substance so they can self administer doses twice daily until their next visit to the study site. Subjects will be instructed to store vials at room temperature and to clean the tip of the spray nozzle with an alcohol wipe after each dose is administered. Vials will be weighted before dispensing and upon return to the clinic 2 wks later to determine how much solution was actually ejected from the vial.

Measurements: A battery of well-validated instruments to quantify psychiatric symptoms, social cognition and social competence will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-IV criteria for paranoid or undifferentiated schizophrenia for at least 1 year.
* Scoring > or equal to 4 on the suspiciousness/persecution (paranoia) subscale of the Positive and Negative Symptoms Scale (PANSS), a full PANSS score > or equal to 60: stability of symptom severity and on the same medication(s) and dose(s) for at least 1 month; low to moderate depressive symptoms.

Exclusion Criteria:

* Low literacy as indicated by an inability to read and understand the consent form.
* Dependence on substances other than tobacco or caffeine.
* Positive urine drug screen for illegal substances or drugs that have not been prescribed.
* Debilitating medical conditions (including AIDS; HIV infection alone will not be grounds for exclusion).
* Major surgery or trauma in the past year will be grounds for exclusion although subjects determined to be recovered and stable may be included at the discretion of the PI.
* Pregnancy, breast-feeding.
* Having given birth in the past 6 months or breast-feeding in the past 3 months.
* Individuals judged unable to learn self-administration of intranasal treatments and/or not sufficiently reliable to do so will be excluded.
* Abnormalities found during medical evaluation will be grounds for exclusion although subjects with laboratory measures barely outside the normal range may be included at the discretion of the Principal Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cort A Pedersen, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Department of Psychiatry — http://www.psychiatry.unc.edu
- See also: UNC Department of Psychiatry Research — http://www.psychiatry.unc.edu/research

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Spray Without Oxytocin: Twice daily intranasal spray without oxytocin (six 0.1 ml insufflations/dose) for 6 weeks.
  nasal spray without oxytocin: 6 insufflations (0.1 metered dose/insufflation) twice daily for 6 weeks
Period: Overall Study
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin
Started | 10 | 7
Completed | 8 | 6
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.88 (7.22) | 35.67 (9.00) | 37.50 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Emotion Recognition as Measured by the Emotion Recognition-40 at the 6 Week Time Point
Description: The Emotion Recognition-40 (ER-40; Kohler, Turner, Gur, & Gur, 2004) consists of a series of 40 faces, shown one at a time on a computer screen. Participants choose the correct emotions based on 5 answer choices: happy, sad, anger, fear and no emotion. Participants indicate the word that best describes the emotion each faces expresses. The stimuli are presented in a randomized order each time they are administered. A scoring program automatically records accuracy and median response time. Range for each emotion (score range) is 0 (no correct responses) to 8 (all faces on each emotion category are correctly identified).
  The ER-40 faces were derived from the University of Pennsylvania Emotion Recognition Task, 96 faces version, and are balanced for equality and intensity of emotion, age, gender and ethnicity.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin
Number analyzed (Participants) | 8 | 6
number of correct responses
  Fear | 7.25 (.89) | 6.67 (1.86)
  Anger | 4.38 (1.30) | 6.17 (1.72)
  Sad | 7.13 (1.46) | 6.50 (1.64)
  Happy | 8.00 (.00) | 7.83 (.41)
  Neutral | 7.25 (.89) | 7.17 (.98)
Statistical Analysis 1: Comparison: Intranasal Spray With Oxytocin; Analysis of fear emotion; Test type: Superiority or Other; p = .61, t-test, 1 sided — Not adjusted for multiple comparisons

2. Secondary Outcome: Clinical Psychiatric Symptoms as Measured by Positive and Negative Syndrome Scale (PANSS) at 6 Weeks
Description: The PANSS consists of 30 items (7 positive psychotic symptoms, 7 negative psychotic symptoms, 16 general psychopathology symptoms) on which subjects are rated (1-7) based upon a semi-standardized interview. Higher scores indicate more/greater symptoms (i.e., greater symptoms of psychosis) and lower scores indicate fewer symptoms (better outcome).
  Possible score range: min, max Total: 30,210 Positive symptoms:7, 49 Negative symptoms:7, 49 General symptoms: 16,112
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: rating on a scale
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin
Number analyzed (Participants) | 8 | 6
rating on a scale
  Positive Symptoms | 14.00 (3.34) | 18.50 (6.22)
  Negative Symptoms | 17.25 (4.20) | 17.17 (3.66)
  General Symptoms | 29.88 (4.91) | 32.67 (4.13)
Statistical Analysis 1: Comparison: Intranasal Spray With Oxytocin; Positive Symptoms; Test type: Superiority; p = 0.008, t-test, 2 sided
Statistical Analysis 2: Comparison: Intranasal Spray With Oxytocin; Negative Symptoms; Test type: Superiority; p = 0.002, t-test, 2 sided
Statistical Analysis 3: Comparison: Intranasal Spray With Oxytocin; General Symptoms; Test type: Superiority; p = 0.04, t-test, 2 sided
Statistical Analysis 4: Comparison: Intranasal Spray Without Oxytocin; Positive Symptoms; Test type: Superiority; p = 0.05, t-test, 2 sided
Statistical Analysis 5: Comparison: Intranasal Spray Without Oxytocin; Negative Symptoms; Test type: Superiority; p = 0.08, t-test, 2 sided
Statistical Analysis 6: Comparison: Intranasal Spray Without Oxytocin; General Symptoms; Test type: Superiority; p = 0.025, t-test, 2 sided

3. Primary Outcome: Theory of Mind as Measured by the Eyes Test at 6 Weeks
Description: The Eyes Test (Baron-Cohen, Wheelwright, Hill, Raste, & Plumb, 2001) consists of 36 photographs where participants are asked to guess the mental state (i.e., what the person is thinking or feeling) from among four choice words. Participants are given a practice item to ensure that they understand the task. Each eye region is displayed on a computer screen with the four choice mental states shown in the four corners of the computer screen (one target word and three foil words). The score range is 0 (no correct responses) to 36 (all stimuli are correctly identified).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin
Number analyzed (Participants) | 8 | 6
correct responses | 22.25 (5.29) | 22.17 (7.83)

4. Primary Outcome: Theory of Mind as Measured by the Brune Test at 6 Weeks
Description: In The Brune Test (Brune, 2003), participants are shown a series of six sets of four cartoon pictures that illustrate interactions between two or more individuals. The cartoon cards were displayed to the participant in a predetermined scrambled order. Participants are asked to rearrange the pictures in an order that conveys a logical story. After the participant arranges the cards, the examiner ensures they are in the correct sequence. If they are not in the correct order, the examiner silently arranges them so they are in the logical sequence.The participant's interpretations of the characters' beliefs are scored as correct or incorrect (zero or one), with higher scores indicating better Theory of Mind. The sum of correct answers is the outcome of interest. The participants can receive a maximum total of 23 points for the questions.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin
Number analyzed (Participants) | 8 | 6
correct responses | 21.13 (1.36) | 22.00 (1.27)
Statistical Analysis 1: Comparison: Intranasal Spray With Oxytocin vs Intranasal Spray Without Oxytocin; Test type: Superiority or Other; p = .03, t-test, 2 sided — Not adjusted for multiple comparisons

5. Primary Outcome: Social Perception as Measured by the Trustworthiness Task at 6 Weeks
Description: The Trustworthiness Task (Adolphs, Tranel, & Damasio, 1998) is comprised of 42 black and white photographs of the faces of unfamiliar people. Participants are shown each picture individually (on a computer monitor) and asked to rate how much they would trust that person (e.g., with their money) on a seven-point scale, ranging from -3 (very untrustworthy) to +3 (very trustworthy). They are provided with a photograph of 0 or an average face (i.e., someone they would neither trust nor distrust) to refer to throughout the task (based on Adolphs et al.'s, 1998 norms). The total score is the sum of the trustworthiness ratings. Possible range is -126 to 126.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: rating on a scale
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin
Number analyzed (Participants) | 8 | 6
rating on a scale | 1.88 (40.98) | 11.33 (34.23)

6. Primary Outcome: Empathy as Measured by the Interpersonal Reactivity Index (IRI) at 6 Weeks
Description: The Interpersonal Reactivity Index (IRI; Davis, 1983) is a self-report measure of cognitive and affective empathy. The IRI consists of 28 items where participants rate how well each item describes them using a five-point scale (1 to 5). The 28 items yield four subscales: perspective taking (PT), empathic concern (EC), fantasy (F), and personal distress (PD). Higher scores indicate a greater empathic response.
  Score range for IRI: min, max Total: 28, 140 PT: 7, 35 EC: 7, 35 F: 7, 35 PD: 7, 35
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: rating on a scale
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin
Number analyzed (Participants) | 5 | 5
rating on a scale
  Total Score | 88.00 (13.71) | 87.00 (8.57)
  Fantasy | 21.60 (4.62) | 26.80 (6.26)
  Emotional Empathy | 23.80 (4.82) | 23.60 (6.88)
  Perspective Taking | 23.40 (2.51) | 19.40 (8.26)
  Distress | 19.20 (4.09) | 17.20 (4.32)
Statistical Analysis 1: Comparison: Intranasal Spray With Oxytocin; IRI-total; Test type: Superiority or Other; p = .784, t-test, 2 sided — Not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Intranasal Spray With Oxytocin; Distress analysis; Test type: Superiority or Other; p = 1.00, t-test, 2 sided
Statistical Analysis 3: Comparison: Intranasal Spray With Oxytocin; Perspective-Taking; Test type: Superiority or Other; p = .03, t-test, 2 sided
Statistical Analysis 4: Comparison: Intranasal Spray With Oxytocin; Emotional empathy analysis; Test type: Superiority or Other; p = .135, t-test, 2 sided
Statistical Analysis 5: Comparison: Intranasal Spray With Oxytocin; Fantasy Analysis; Test type: Superiority or Other; p = .681, t-test, 2 sided
Statistical Analysis 6: Comparison: Intranasal Spray Without Oxytocin; Distress analysis; Test type: Superiority or Other; p = 1.00, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Intranasal Spray With Oxytocin | Intranasal Spray Without Oxytocin
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 1/10 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Spray With Oxytocin (N=10) | Intranasal Spray Without Oxytocin (N=7)
Serious Adverse Events (Psychiatric disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Spray With Oxytocin (N=10) | Intranasal Spray Without Oxytocin (N=7)
low blood pressure due to blood-draw (Vascular disorders) | 1 (1) | 0 (0) — This subject experienced a drop in blood pressure (79/43) and heart rate (46) during the blood draw for the baseline visit. Subject was given breakfast and felt better after a few minutes and blood pressure/heart rate returned to normal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No